CLINICAL TRIAL: NCT06205394
Title: Improving the Breast Cancer Care Delivery Model for Sex and Gender Minority Survivors (Intended for SGM)
Brief Title: Improving The Breast Cancer Care Delivery Model for Sex and Gender Minority Survivors, Intended for SGM Study
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Arthur, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-22123; NCI-2023-00667 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-22123 (Other: Ohio State University Comprehensive Cancer Center)
Record Dates: First submitted 2023-10-31; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP 1 (focus group): Cancer survivors participate in a focus group on study.
  Interventions: Other: Non-Interventional Study
- GROUP 2 (interview): Breast cancer clinicians undergo a semi-structured interview on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates Improving the Breast Cancer Care Delivery Model for Sex and Gender Minority (INTENDED for SGM) in identifying the patient, support person and provider barriers to quality care in SGM breast/chest cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the important ways the iCanDecide breast cancer decision aid needs revised for SGM people, and how best to integrate a culturally-relevant tool into clinical practice.

OUTLINE: This is an observational study.

AIM 1: Interview transcripts from SANGRIA study utilized to explore the values, preferences and key considerations for breast cancer treatment decision making in SGM individuals.

AIM 2: Patients are assigned to 1 of 2 groups.

GROUP 1: Cancer survivors participate in a focus group on study.

GROUP 2: Breast cancer clinicians undergo a semi-structured interview on study.

ELIGIBILITY:
Inclusion Criteria:

* SURVIVORS:

  * Self-identify as a member of the sex and gender minority community or partner with an individual of the same sex or gender
  * Must be a breast cancer survivor, in active treatment or completed active treatment in the last 10 years (not including hormone therapy)
  * Be over age 18
  * English-speaking
  * Received care in the US

BREAST ONCOLOGY CLINICIANS: Physicians, advanced practice providers, nurses, psychologists and social workers will be eligible if they:

* Provide care and/or surgical decision support to individuals diagnosed with early stage breast cancer in the US
* Are English-speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer survivors that self-identify as a member of the sex and gender minority community or partner with an individual of the same sex or gender and breast oncology clinicians recruited through Ohio State University Comprehensive Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Survivor participant feedback, opinions, and preferences for breast cancer care | At completion of study up to 2 years
  Data is verbally reported and collected in focus groups
Clinician participant reports of experiences, opinions, and knowledge of caring for LGBTQ+ people | At completion of study up to 2 years
  Data is verbally reported and collected in interviews

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Arthur, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Informed Consent Form: Patients (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT06205394/ICF_000.pdf
  • Informed Consent Form: Clincians (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT06205394/ICF_001.pdf